CLINICAL TRIAL: NCT07279116
Title: Phase 1 Trial of ABY-029 Fluorescence in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: ABY-029 Head & Neck Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph A. Paydarfar, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02002698; R01CA167413 (NIH)
Record Dates: First submitted 2025-12-08; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: ABY-029; Affibody; Molecular Fluorescence-Guided Surgery; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — ABY-029

STUDY DESIGN:
Intervention Model Description: Twelve (12) participants with likely EGFR-positive tumors will be enrolled, alternating between two ABY-029 administration doses (the 6X dose and 10X dose), until a total of 24 participants have been enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABY-029 6X dose group (Experimental): ABY-029 will be administered at the 6X dose level prior to surgery to participants with HNSCC.
  To understand the safety of ABY-029, investigators will collect blood samples before and after surgery at these time points: before the drug is given to the participant, one or two minutes after participants are given the drug, about 15 minutes after participants are given the drug, and just prior to anesthesia. Investigators will also collect one urine sample and take EKG readings to monitor the participant's heart before surgery. Investigators will repeat blood, urine and EKG tests when participants are in the hospital after surgery.
  Interventions: Drug: ABY-029
- ABY-029 10X dose group (Experimental): ABY-029 will be administered at the 10X dose level prior to surgery to participants with HNSCC.
  To understand the safety of ABY-029, investigators will collect blood samples before and after surgery at these time points: before the drug is given to the participant, one or two minutes after participants are given the drug, about 15 minutes after participants are given the drug, and just prior to anesthesia. Investigators will also collect one urine sample and take EKG readings to monitor the participant's heart before surgery. Investigators will repeat blood, urine and EKG tests when participants are in the hospital after surgery.
  Interventions: Drug: ABY-029

INTERVENTIONS:
Drug: ABY-029 — ABY-029 will be administered via single intravenous injection to subjects with HNSCC approximately 1-3 hours prior to surgery.
  All research procedures will occur during surgery. The research procedures involve image and measurement data collection and biopsy specimen sampling. Research data collection will occur at 3 or 4 time points during surgery using either standard-of-care tools and methods or non-significant risk experimental devices.
  No follow-up visit will be required of participants. Participants will be monitored for possible adverse events for approximately 30 days by the operating surgeon involved in the clinical trial procedures and through review of participant medical records.

SUMMARY:
The purposes of the research trial are to study the safety of ABY-029 and to understand how much of the drug is needed to reach head and neck squamous cell carcinomas (HNSCC) so it can be visualized best by surgeons. Investigators will do this by comparing two groups of participants that receive different, very small amounts of ABY-029. Investigators will use an imaging system during surgery to record the amount of ABY-029 in the participant's tumor and in the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis of head and neck squamous cell carcinoma with planned surgical resection of the oral cavity, oropharynx, larynx, or hypopharynx.
2. Tumor judged to be operable.
3. Valid informed consent by participant.
4. Age ≥ 18 years old.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with a medical history of (Grade 2 or higher) hepatic/renal function compromise.
2. Prisoners
3. Individuals who are pregnant or breast feeding.
4. Patients on experimental or approved anti-EGFR targeted therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to ABY-029 | one month
  To study the safety of ABY-029, adverse events related to 6X and 10X doses of ABY-029 will be tracked following surgery, and the proportion of study-drug related adverse events at 6X and 10X doses will be compared statistically for significant differences.
Diagnostic accuracy of measured ABY-029 fluorescence ex-vivo in surgical specimens | up to three months
  To measure the diagnostic performance of ABY-029, the diagnostic accuracy of measured ABY-029 fluorescence ex-vivo in surgical specimens histologically confirmed as tumor from participants receiving the 6X microdose and 10X microdose.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Paydarfar, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: No